CLINICAL TRIAL: NCT07089550
Title: PSMA PET for Treatment Response evaLuation of systemIC Therapies in prostAte caNcer (PELICAN), an Italian Multicenter Study
Brief Title: PSMA PET for Treatment Response evaLuation of systemIC Therapies in prostAte caNcer (PELICAN)
Acronym: PELICAN
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Collaborators: Ospedale Policlinico San Martino (Other); Ospedale Santa Croce-Carle Cuneo (Other); Azienda Ospedaliera Universitaria Policlinico "G. Martino" (Other)
Responsible Party: Principal Investigator, Andrea Farolfi, MD, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Other Study IDs: 737/2024/Oss/AOUBO
Record Dates: First submitted 2025-05-28; First posted 2025-07-28 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: PSMA Positive Tumors or Tumor Tissues; Prostate Cancer Metastatic
Keywords: PSMA PET/CT; mCRPC; mHSPC

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- PELICAN population: Patients with either hormone-sensitive (HSPC) or castration-resistant (CRPC) prostate cancer
  Interventions: Radiation: PSMA PET/CT scan

INTERVENTIONS:
Radiation: PSMA PET/CT scan — All Patients undergoing PSMA PET for pre-treatment disease staging with different radiotracers ([68Ga]Ga-PSMA-11, [18F]-DCFPyL, [18F]-PSMA-1007).

SUMMARY:
This prospective clinical study aims to evaluate the predictive power of PSMA PET imaging in patients with advanced prostate cancer who are receiving systemic drug therapies.

The primary goal is to identify prognostic factors derived from PSMA PET imaging. These factors include the number of cancer lesions, the size of the tumor, and measurements known as SUVmax and SUVmean. By identifying these factors, the investigators aim to better group patients and predict those who may have a less favorable outcome. While PSMA PET imaging is highly accurate in locating cancer sites within the body, its ability to predict treatment response has not yet been thoroughly studied in a prospective manner for this patient population.

This study will assess the predictive role of PSMA PET imaging and its ability to forecast treatment response across a range of systemic therapies, including hormone therapy and chemotherapy, in patients with both hormone-sensitive (HSPC) and castration-resistant (CRPC) prostate cancer.

DETAILED DESCRIPTION:
Purpose: to determine the prognostic value of PSMA PET imaging in patients diagnosed with advanced prostate cancer who are undergoing systemic therapies. The study will enroll patients with either hormone-sensitive (HSPC) or castration-resistant (CRPC) disease.

Design of the register: observational, pharmacological, non-profit, prospective, multicentric.

Duration of the record: The expected duration for the collection of PET/CT-PSMA examinations is 9 years.

The primary objective is to evaluate the predictive capacity of PSMA PET, focusing on quantitative parameters such as the number of lesions, tumor volume (as assessed by metabolic tumor volume - MTV), maximum standardized uptake value (SUVmax), and mean standardized uptake value (SUVmean), to stratify patient risk and predict unfavorable clinical outcomes (e.g., progression-free survival, overall survival).

This research will address the existing knowledge gap regarding the predictive ability of PSMA PET beyond its established role in disease localization. Specifically, the study will investigate if PSMA PET parameters can forecast response to a spectrum of systemic treatments, including but not limited to: abiraterone, enzalutamide, apalutamide, darolutamide, docetaxel, cabazitaxel, olaparib, radiotherapy, 177-lutetium PSMA, and 225-actinium PSMA.

Secondary objectives include:

* Identifying PSMA PET-derived biomarkers that predict response to the aforementioned systemic therapies.
* Assessing the incremental prognostic and predictive value of PSMA PET in conjunction with standard imaging modalities, namely CT, MRI, and bone scan, in patients undergoing multiple imaging assessments.
* Evaluating the correlation between changes in PSMA PET-derived tumor volume during treatment and clinical outcomes.

This study will leverage quantitative imaging data obtained from PSMA PET to develop predictive models that may refine patient stratification and personalize treatment strategies for advanced prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of advanced prostate cancer (excluding neuroendocrine carcinoma);
* Patients undergoing PSMA PET for pre-treatment disease staging;
* Candidates to receive one or more of the following systemic therapies, in combination or alone: abiraterone, enzalutamide, apalutamide, darolutamide, docetaxel, cabazitaxel, olaparib, radiotherapy, lutetium-177-PSMA, actinium-225-PSMA;
* Provision of signed informed consent for study participation and data handling.

Exclusion Criteria:

* Inability to remain supine and still for the PET/CT image acquisition;
* Prostate cancer with a known significant neuroendocrine component;
* Presence of another concurrent malignancy, with the exception of non-melanoma skin cancer.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: This study will enroll male patients aged 18 years or older with a histologically confirmed diagnosis of advanced prostate cancer (excluding neuroendocrine carcinoma).
Sampling Method: Non-Probability Sample
Enrollment: 1300 (Estimated)
Dates: Start 2025-04-02 (Actual); Primary Completion 2034-04-26 (Estimated); Study Completion 2034-04-26 (Estimated)

PRIMARY OUTCOMES:
number of PSMA-avid lesions (count) | From baseline PET/CT through study completion, an average of 2 years
  number of PSMA-avid lesions (count)
metabolic tumor volume (MTV in cm 3) | From baseline PET/CT through study completion, an average of 2 years
  metabolic tumor volume (MTV in cm 3)
maximum standardized uptake value (SUVmax, dimensionless) | From baseline PET/CT through study completion, an average of 2 years
  maximum standardized uptake value (SUVmax, dimensionless)
mean standardized uptake value (SUVmean, dimensionless) | From baseline PET/CT through study completion, an average of 2 years
  mean standardized uptake value (SUVmean, dimensionless)

SECONDARY OUTCOMES:
Prediction of Treatment Response via PSMA PET | From baseline PET/CT through study completion, an average of 2 years
  Predictive value of PSMA PET-derived parameters in forecasting patient response to systemic therapies (abiraterone, enzalutamide, apalutamide, darolutamide, docetaxel, cabazitaxel, olaparib, radiotherapy, 177-lutetium PSMA, 225-actinium PSMA). This will be assessed by correlating PSMA PET metrics with established clinical and radiological response criteria for each respective therapy.
Comparative Analysis of Imaging Modalities | From baseline PET/CT through study completion, an average of 2 years
  Incremental predictive and prognostic value of PSMA PET, when used in conjunction with standard imaging techniques (CT, MRI, bone scan). This will involve comparing the predictive accuracy of PSMA PET alone versus combined imaging approaches in predicting treatment outcomes and patient survival.
Assessment of Tumor Volume Dynamics | From baseline PET/CT through study completion, an average of 2 years
  Correlation between changes in PSMA PET-derived tumor volume (MTV) during the course of systemic treatment and patient clinical outcomes, including but not limited to, progression-free survival and overall survival. This will assess the utility of dynamic MTV changes as a surrogate marker for treatment response.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Farolfi, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (4):
- Italy (4):
  - Nuclear Medicine, IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy
  - Azienda Ospedaliera Santa Croce e Carle - ospedale Santa Croce, Cuneo, Italy
  - U.O. Medicina Nucleare, IRCCS Ospedale Policlinico San Martino, Genova, Italy
  - UOC Medicina Nucleare, AOU Policlinico G.Martino, Messina, Italy

IPD SHARING:
Plan to Share IPD: Undecided